CLINICAL TRIAL: NCT03075046
Title: Use of 405nm Blue Light Emitting Diode in the Treatment of Women With Vulvovaginal Candidiasis: a Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Collaborators: Vitale SG M.D. (Unknown); University of Messina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CentroAAP
Record Dates: First submitted 2017-02-22; First posted 2017-03-09 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Candidiasis, Vulvovaginal
Keywords: Blue Light Emitting Diode; Women
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- blue LED 405 nm in vulvovaginal candidiasis (Experimental): It will be applied the a 405 nm blue LED in a closed room by a physiotherapist for 30 minutes. The apparatus shall be supported on a tripod, statically, externally, 5 cm away from the vulva and vagina region, with the patient naked, in gynecological stretcher and lithotomy position. The protocol will consist of only one session. This part of the study will see if there is fungicidal effect of the blue led 405 nm
  Interventions: Device: Blue LED 405 nm; Other: Questionnaire of anamnesis
- blue LED 405 nm in healthy women (Experimental): It will be applied the a 405 nm blue LED in a closed room by a physiotherapist for 30 minutes. The apparatus shall be supported on a tripod, statically, externally, 5 cm away from the vulva and vagina region, with the patient naked, in gynecological stretcher and lithotomy position. The protocol will consist of only one session.This part of the study will see the security and the effects of the blue led 405 nm in healthy vaginal microflora
  Interventions: Device: Blue LED 405 nm; Other: Questionnaire of anamnesis
- Sociodemographic data of women with vulvovaginal candidiasis (No Intervention): The women will answer some questions of the anamnesis as: Age, weight, height, form of intimate hygiene, and others to evaluate possible correlations of these data with the presence of vulvovaginal candidiasis

INTERVENTIONS:
Device: Blue LED 405 nm — It will be applied a 405 nm blue Tonderm LED with a power of 1.66 W / m2, in a closed room by a physiotherapist for 30 minutes. The apparatus shall be supported on a tripod, statically, externally, 5 cm away from the vulva and vagina region, with the patient naked, in gynecological stretcher and lithotomy position. The protocol will consist of only one session.
  Arms: blue LED 405 nm in healthy women; blue LED 405 nm in vulvovaginal candidiasis
Other: Questionnaire of anamnesis — The participants will answer the anamnesis Questionnaire that will be applied by the physiotherapist
  Arms: blue LED 405 nm in healthy women; blue LED 405 nm in vulvovaginal candidiasis

SUMMARY:
Vulvovaginal candidiasis (CVV) is an infectious process of the female genitourinary tract, an important health issue due to the high incidence and difficulties encountered in the treatment. Therefore, new therapeutic modalities are sought with the capacity to minimize drug side-effects and to reduce recurrent cases. The objective of this stufy is to evaluate the clinical and microbiological response of the 405 nm blue light emitting diode in the treatment of women with vulvovaginal candidiasis and in women with healthy gentourine treatment. A clinical trial was conducted involving 40 women, divided into two groups, the first group consisting of women with a confirmed CVV diagnosis and a second group formed by women with a healthy genitourinary tract, without symptoms and symptoms of the disease. Both groups underwent clinical evaluation and examination with endocervice collection with gynecologist before and after a session of application of the Blue Light Emitting Diode of 405 nm, lasting 4.5 minutes. There will also be an evaluation of the effects of the diary through the questionnaire answered before and after the participants' treatment. It is expected that the 405 nm blue LED will destroy the CVV fungus demonstrated by laboratory examination and also improve the signs and results analyzed by the gynecologist and participants.

DETAILED DESCRIPTION:
A current treatmente proposal is the use of blue LED of 405 nm wich is a light that has antimicrobial effect when exposed to endogenous porphyrin of the pathogens. This exposition produces reactive oxigen and it causes cells death with no possibilities of resistance by the fungus.

ELIGIBILITY:
Inclusion Criteria:

* women betwen 18 and 65 years old, with clinical suspect of vulvovaginal candidiasis and with health vaginal tract

Exclusion Criteria:

* Women with pacemakers, with diagnosis and / or suspicion of neoplasias, cognitive deficits, neurological and / or psychiatric diseases, pregnant women and women who have used oral antibiotics, fungicides, corticosteroids and vaginal creams in the last 30 days

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Description of types of cells done by oncology and microflora cytology in women treated by blue light emitting diode | 15 days
  These exam will be done by the collect of vaginal secretion to analyse types of cells and organisms
Amount of clue cells quantified by fresh citology in vaginal secretion of women treated by blue light emitting diode | 5 hours
  These exam will be done by the collect of vaginal secretion using KOH 10% to analyse clue cells by percentage %
Value of vaginal pH measurement in women treated by blue light emitting diode | 30 minutes
  These exam will be done by the collect of vaginal secretion using a ph measuring tape to analyse the hydrogen potential in -log10 [aH+] in women treated by blue light emitting diode. It will be used the numeric scale of pH value
Quantification of fungal colony units by the fungus culture in vaginal secretion of women treated by blue light emitting diode | 15 days
  These exam will be done by the collect of vaginal secretion using Colony Forming Unit CFU in women treated by blue light emitting diode

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pereira E Silva ACM, Brito MB, Robatto M, Pavie MC, Villas Boas AQ, Sousa R, Lordelo P. Blue Light-Emitting Diode Therapy for Chronic Vulvovaginitis Symptoms: A Series of Cases. Photobiomodul Photomed Laser Surg. 2022 Nov;40(11):747-750. doi: 10.1089/photob.2022.0038. PMID 36395084
- [Derived] Pavie MC, Robatto M, Bastos M, Tozetto S, Boas AV, Vitale SG, Lordelo P. Blue light-emitting diode in healthy vaginal mucosa-a new therapeutic possibility. Lasers Med Sci. 2019 Jul;34(5):921-927. doi: 10.1007/s10103-018-2678-3. Epub 2018 Nov 7. PMID 30406341
- Available data/document: Informed Consent Form — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf